CLINICAL TRIAL: NCT02668354
Title: Cancer in Infants: South Egypt Cancer Institute Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Cancer in Infants SECI
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Infantile Neoplasms
Keywords: Childhood Cancer; Pediatric Oncology; Infant tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate the spectrum of various types of malignant neoplasms of infancy, according to the experience of South Egypt Cancer Institute, which represents the largest referral site in Upper Egypt.

DETAILED DESCRIPTION:
Background:

Cancer in the first year of life is relatively rare ; however, the age of peak cancer incidence among children occurs during the first year of life, representing 10% of all cancer that was diagnosed among children younger than 15 years of age. Female and male infants have essentially the same overall cancer incidence rates.

Cancer occurring in infants often has a clinical and biological behavior that is different from cancers occurring in older children. The histologic distribution of cancers in infants and that in older children are also different.

Patients & Methods:

From January 2001 to December 2015, retrieval & analysis of the medical records of infant patients, diagnosed with any of malignant tumors, at the pediatric oncology department at South Egypt Cancer Institute will be done. Pathologic diagnoses & age of the patients will be verified for the enrollment in the study. The collected data will be analyzed to delineate the spectrum of these disease entities, their clinico-pathologic features, associated patients' demographics and characteristics, treatment modalities received, and outcomes of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than or equal to 1 year.
* Patients diagnosed with any of malignant neoplasms.

Exclusion Criteria:

• Patients whose age more than 1 year.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants, those diagnosed with any of malignant neoplasms, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Chen, S.-H., Y.-L. Liu, et al. (2014). Infants with cancer: A unique population. Journal of Experimental & Clinical Medicine 6(1): 1-9.
- [Background] Dreyer, Z., D. Indelicato, et al. (2011). Infants and adolescents with cancer: special considerations. In: Pizzo PA, Polackand DG, editors. Principles and practice of pediatric oncology. 6th ed. Riverwoods, IL: Lippincott Williams & Wilkins.
- [Background] Gurney, J. G., M. A. Smith, et al. (1999). Cancer among infants. Cancer incidence and survival among children and adolescents: United States SEER Program 1975-1995: 149-156.
- [Background] Yang CP, Hung IJ, Jaing TH, Shih LY, Chang WH. Cancer in infants: a review of 82 cases. Pediatr Hematol Oncol. 2005 Sep;22(6):463-81. doi: 10.1080/08880010591002233. PMID 16169813